CLINICAL TRIAL: NCT07253896
Title: Efficacy and Safety of AK104 Combined With Chemotherapy and Cetuximab or Bevacizumab as Second-line Treatment in MSS Type Metastatic Colorectal Cancer Based on RAS Gene Status
Brief Title: Efficacy and Safety of AK104 Combined With Chemotherapy and Cetuximab or Bevacizumab
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Ying Yuan, MD, Second Affiliated Hospital, School of Medicine, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IR2023176
Record Dates: First submitted 2024-01-29; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Safety
Keywords: colorectal cancer; AK104; chemotherapy; cetuximab; bevacizumab
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK104 Combined With Chemotherapy and Cetuximab or Bevacizumab (Experimental): AK104 Combined With Chemotherapy and Cetuximab or Bevacizumab
  Interventions: Drug: AK104 and cetuximab or bevacizumab and FOLFIRI

INTERVENTIONS:
Drug: AK104 and cetuximab or bevacizumab and FOLFIRI — AK104 and cetuximab or bevacizumab and FOLFIRI as the second line

SUMMARY:
Evaluate the objective response rate (ORR) of AK104 combined with chemotherapy and cetuximab or bevacizumab in second-line treatment of MSS type advanced colorectal cancer

DETAILED DESCRIPTION:
This study is a single arm, open label, single center clinical study aimed at evaluating the efficacy and safety of candenizumab combined with chemotherapy and targeted drugs (cetuximab or bevacizumab) in second-line treatment of MSS type advanced metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. Voluntarily sign a written ICF. 2. Age at enrollment: ≥ 18 years old, ≤ 75 years old, both male and female. 3. The Eastern Cancer Collaborative Organization (ECOG) has a physical fitness score of 0 or 1.

  4. The expected survival period is ≥ 3 months. 5. Metastatic colorectal adenocarcinoma confirmed by histology or cytology. 6. Microsatellite instability (MSI) status is MSI-L or MSS type human. 7. The metastatic lesion cannot be removed and is not suitable for curative surgical treatment.

  8. Previously only received first-line systemic anti-tumor therapy based on oxaliplatin (FOLFOX or CAPOX), and other systemic anti-tumor treatments for metastatic colorectal cancer are not allowed. Note: For subjects who have previously received neoadjuvant therapy, adjuvant therapy, or curative radiotherapy and chemotherapy, if disease progression occurs during or within 6 months after treatment, it is considered that they have received first-line treatment.

According to RECIST v1.1, subjects must have at least one measurable lesion. For subjects who have previously received radiotherapy, if there are no other lesions that can be selected as target lesions and there is objective evidence of significant progression after radiotherapy, the irradiated lesions can be considered as target lesions.

10. The subjects are required to provide 15 recently archived or freshly obtained FFPE pathological sections of tumor tissue.

11. Determine good organ function through the following requirements:

a) Hematology (no use of any blood components or cell growth factor branches within 7 days prior to starting treatment)

Holding treatment:

i. Neutrophil absolute value ANC ≥ 1.5 × 109/L (1500/mm3); Ii. Platelet count ≥ 100 × 109/L (100000/mm3); Iii. Hemoglobin ≥ 90 g/L. b) Kidney: i. The calculated value of creatinine clearance rate * (CrCl) is ≥ 50 mL/min

*The Cockcroft Fault formula will be used to calculate CrCl (Cockcroft Fault formula) CrCl (mL/min)={(140- age) × Weight (kg) × F} /(SCr (mg/dL) × 72) F=1 for males; F=0.85 for women; SCr=serum creatinine. Ii Urinary protein ≤ 1+or 24-hour (h) urinary protein quantification<1.0 g. c) Liver: i. Total serum bilirubin (TBil) ≤ 1.5 × ULN; For liver metastasis or evidence to confirm/suspect Subjects with Gilbert disease, TBil ≤ 3 × ULN Ii. AST and ALT ≤ 2.5 × ULN; For subjects with liver metastasis, AST and ALT ≤ 5 × ULN Iii. Serum albumin (ALB) ≥ 28 g/L d) Coagulation function: i. International Standardization Ratio

Exclusion Criteria:

* 1. Patients with known MSI-H or dMMR. 2. Patients with BRAF mutations. 3. Subjects suffered from other malignant tumors within 3 years before enrollment, except for cured local tumors (such as basal cell skin cancer, squamous cell skin cancer, superficial bladder cancer, cervical carcinoma in situ, etc.).

  4. Simultaneously enroll in another clinical study, unless it is an observational, non-interference clinical study or a follow-up period of an intervention study.

  5. Have received any immunotherapy against tumors in the past, including immune checkpoint inhibitors (such as anti-PD-1 antibodies, anti-PD-L1 antibodies, anti-CTLA-4 antibodies, etc.), immune checkpoint agonists (such as ICOS, CD40, CD137, GITR, OX40 antibodies, etc.), immune cell therapy, and any treatment targeting the immune mechanism of tumors.

  6. Patients with active autoimmune diseases that require systematic treatment within the past two years (such as using medication to improve the condition, corticosteroids, immunosuppressive agents), and replacement therapy (such as thyroid hormone, insulin, or physiological corticosteroid replacement therapy for adrenal or pituitary dysfunction) are not considered as systematic treatment.

  7. A history of active or previous inflammatory bowel disease (such as Crohn's disease, ulcerative colitis, or chronic diarrhea).

  8. History of immunodeficiency; HIV antibody test positive individuals; Currently using systemic corticosteroids or other immunosuppressants for a long time.

  9. Subjects who are known to have active pulmonary tuberculosis (TB) and suspected to have active TB need to undergo clinical examination to exclude them; Known active syphilis infection.

  10. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.

  11. Previous or current non infectious pneumonia/interstitial lung disease requiring systemic glucocorticoid treatment.

  12. Severe infections occurring within 4 weeks prior to the first administration, including but not limited to comorbidities requiring hospitalization, sepsis, or severe pneumonia; Active infections that have received systemic anti infective treatment within two weeks prior to the first administration (excluding antiviral treatment for hepatitis B or C).

  13. Subjects with active hepatitis B (HBsAg positive and HBV-DNA exceeding 1000 copies/ml (200 IU/ml) or above the lower detection limit, whichever is higher). Note: Non active or asymptomatic carriers, treated and stable hepatitis B subjects with HBV DNA ≤ 1000 IU/mL are eligible for inclusion. Subjects with hepatitis B are required to receive anti hepatitis B virus treatment during the study treatment.

  14. Active hepatitis C subjects (HCV antibody positive and HCV RNA levels above the detection limit).

  15. Those who have undergone major surgical procedures or experienced severe trauma within 30 days prior to the first administration, or have planned major surgical procedures within 30 days after the first administration (as determined by the investigator); Minor local surgery performed within 3 days prior to initial administration (excluding peripheral venous puncture and central venous catheterization and intravenous infusion port implantation)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2026-01-03 (Estimated); Study Completion 2027-01-03 (Estimated)

PRIMARY OUTCOMES:
objective response rate | the proportion of lung cancer patients participating in clinical research who, after receiving treatment, achieve a significant reduction in tumor volume
  The proportion of patients whose tumor volume has decreased by 30% and can be maintained for more than 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ying Yuan, Dr, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (2):
- China (2):
  - the Second Affiliated Hospital of Medical College of Zhejiang University, Hangzhou, Zhejiang
  - the Second Affiliated Hospital of Medical College of Zhejiang University, Hangzhou

IPD SHARING:
Plan to Share IPD: No